CLINICAL TRIAL: NCT03758846
Title: Comparing Conventional and Alternative Therapies for Improving Motor Impairment, Fall-risk and Overall Physical Function
Brief Title: Alternative Therapies for Improving Motor Impairment, Fall-risk and Overall Physical Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Tanvi Bhatt, Associate Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2012-0111; 2P30AG022849-11 (NIH)
Record Dates: First submitted 2018-11-21; First posted 2018-11-29 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Chronic Stroke; Healthy Aging
Keywords: Dual-task training; Cognitive-motor training; Conventional training; Virtual-reality exergaming; Dance Therapy
MeSH Terms: interventions — Dance Therapy; Aging

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cognitive-motor Exergaming (Experimental): A total of 6 Wii-fit games: Bubble balance, Table Tilt, Tightrope walking, Soccer head, Basic Run and Basic Step. A total of 6 cognitive tasks namely Digit recall, repeated letter, word list generation (category and alphabets), mental arithmetic, analogies. Each session was divided into 3 sub-sessions. Every Wii-fit game was played with any 3 cognitive tasks. The combination of games with cognitive tasks was randomized in such a manner that all the cognitive tasks were played with the Wii-fit games in that session. Breaks were provided after each sub-session or when the participant demanded one or when the research personnel noticed any discomfort of the participant.
  Interventions: Behavioral: Cognitive-motor exergaming
- Conventional balance Training for people with Chronic stroke (Active Comparator): The sessions were divided into 10 minutes of warm-up that involved active movements of the body (arm movements, trunk twists, lunges). Next 15 minutes consisted of functional strengthening exercises like high stepping, lunges, squats, resistance training using therabands and weights. Following 35 minutes included balance training exercises like one leg standing, tandem standing, sit to stand exercises, reach outs and step-ups. Last 10-15 minutes were spent treadmill walking. Breaks were provided in between the exercise training as and when needed by the participant.
  Interventions: Behavioral: Conventional balance Training
- Dance Therapy for Stroke (Experimental): Virtual-reality based dance training - Participants received Virtual-reality based dance training for 6 weeks using the commercially available Kinect dance game (Microsoft Inc., Redmond, WA, U.S.A.) "Just Dance 3". The six week session consisted of 5 sessions/week, next two weeks of 3 sessions/week and last two weeks of 2 sessions/week, for a total of 20 sessions. Participants played on 10 songs for the first 2 weeks, progressing to 12 songs during the 3nd and 4th weeks with an addition of 2 more songs of their choice during the last two weeks. Participants played on alternating slow- and fast-paced songs (each maximum of 4 minutes in duration) with a five minutes break after a set of one slow and fast song.
  Interventions: Behavioral: Dance Therapy for Stroke
- Dance Therapy for Older Adults (Experimental): Virtual-reality based dance training - Participants received Virtual-reality based dance training for 6 weeks using the commercially available Kinect dance game (Microsoft Inc., Redmond, WA, U.S.A.) "Just Dance 3". The six week session consisted of 5 sessions/week, next two weeks of 3 sessions/week and last two weeks of 2 sessions/week, for a total of 20 sessions. Participants played on 10 songs for the first 2 weeks, progressing to 12 songs during the 3nd and 4th weeks with an addition of 2 more songs of their choice during the last two weeks. Participants played on alternating slow- and fast-paced songs (each maximum of 4 minutes in duration) with a five minutes break after a set of one slow and fast song.
  Interventions: Behavioral: Dance Therapy for Older adults
- Conventional therapy - Home education for Older adults (Active Comparator): Participants received a one-hour education on conventional physical exercises and fall prevention.
  Interventions: Behavioral: Home education for Older adults

INTERVENTIONS:
Behavioral: Cognitive-motor exergaming — Participants undergo 6 weeks of cognitive-motor exergaming using Wii-fit Nintendo. The 6 weeks included a total of 20 session distributed in the following manner: 5 sessions/week for 1-2 week, 3 session/week for 3-4 week, 2 sessions/week for 5-6 week. Each session lasted for about 90 minutes with rests included.
  Other Names: Dual-task training; Wii-fit exergaming; Virtual-reality training
  Arms: Cognitive-motor Exergaming
Behavioral: Conventional balance Training — Participants undergo 6 weeks of conventional exercise training. The 6 weeks included a total of 20 session distributed in the following manner: 5 sessions/week for 1-2 week, 3 session/week for 3-4 week, 2 sessions/week for 5-6 week. Each session lasted for about 90 minutes with rests included.
  Other Names: Balance training
  Arms: Conventional balance Training for people with Chronic stroke
Behavioral: Dance Therapy for Stroke — Participants will receive therapy using the "Just Dance" using the commercially available Kinect gaming system (Microsoft Inc, Redmond, WA, USA. Each song involves repetitive action for each dance step (at least 20 repetitions over the entire song) and visual cues on the screen (a stick figure at the bottom right) indicating the upcoming dance step. Participant's playing the game to reduce risk of exercise related adverse effects. Participants will dance on 10 songs starting from a slow-pace progressing to a medium pace (each max 5 minutes long). Participants will receive 5 minutes rest after playing on each song. This will be conducted by two physical therapists.
  Other Names: Exergaming-based dance
  Arms: Dance Therapy for Stroke
Behavioral: Dance Therapy for Older adults — Participants will receive therapy using the "Just Dance" using the commercially available Kinect gaming system (Microsoft Inc, Redmond, WA, USA. Each song involves repetitive action for each dance step (at least 20 repetitions over the entire song) and visual cues on the screen (a stick figure at the bottom right) indicating the upcoming dance step. Participant's playing the game to reduce risk of exercise related adverse effects. Participants will dance on 10 songs starting from a slow-pace progressing to a medium pace (each max 5 minutes long). Participants will receive 5 minutes rest after playing on each song. This will be conducted by two therapists.
  Other Names: Exergaming-based dance
  Arms: Dance Therapy for Older Adults
Behavioral: Home education for Older adults — Participants will receive a one-hour education on conventional physical exercises.
  Other Names: Fall prevention
  Arms: Conventional therapy - Home education for Older adults

SUMMARY:
Neurological impairment such as stroke and aging is a leading cause of adult disability. Traditional rehabilitative therapies can help regain motor function and ameliorate disability. There are increasing community and other facilities offering rehabilitation in the form of conventional, recreational and alternative (Yoga, Tai-chi) therapy. However, the implementation of these conventional therapy techniques in individuals with a neurological disorder like stroke and the elderly population is tedious, resource-intensive, and costly, often requiring transportation of patients to specialized facilities. Based on recent evidence suggesting significant benefits of repetitive, task-orientated training, investigators propose to evaluate the feasibility of an alternative therapies such as exergaming based therapy to improve overall physical function of community-dwelling individuals with neurological impairments and the elderly, compared to conventional therapeutic rehabilitation. This pilot study aims to systematically obtain pilot data on compliance and efficacy as well as performing power analysis and sample size calculation for developing it into a randomized controlled trial for extramural funding purposes. The objective of the study is to determine the safety, feasibility, compliance and efficacy of exergaming therapy to improve overall physical function of community-dwelling chronic stroke individuals and the elderly population.

DETAILED DESCRIPTION:
While conventional balance training facilitates balance control and gait functions, the exercises involved in the training are labor-intensive, highly repetitious leading to monotonicity and decreased motivation levels. Therefore, many health care researchers are involved in identifying various methods to reduce the risk of falls addressing the barriers in conventional training methods while having the potential to translate it at home. A pilot study identified that supplementary cognitive training along with Wii-fit balance training resulted in improving dual-task volitional balance control post-stroke. Based on this preliminary finding, this current pilot study aimed to identify:

1. The efficacy of cognitive-motor exergaming (with Wii-fit) compared to conventional balance training among people with chronic stroke
2. Exergaming (with Kinect) on domains of balance control and cognition among people with chronic stroke
3. The efficacy of Exergaming (with Kinect) compared to conventional balance training method on domains of balance control and cognition among healthy older adults

This pilot study used Wii-fit Nintendo/ Microsoft Kinect, an off the shelf, commercially available and a cost-effective device that provides similar benefits of exergaming. Community-dwelling people with chronic stroke and healthy older adults involved in the study underwent 6 weeks of exergaming or conventional balance training in a tapering manner in a laboratory setting. Participants were assessed for motor and cognitive performance in the laboratory during volitional and reactive balance control while performing a secondary cognitive task. The performance outcome determined the effect on cognitive-motor interference during dual-tasking.

ELIGIBILITY:
Inclusion/Exclusion criteria for Stroke

Inclusion Criteria:

* Participants should be 18 to 90 years of age.
* Presence of Chronic stroke (onset of stroke more than six months) confirmed by a physician
* Ability to stand independently for 5 minutes without an assistive device or any physical assistance
* Ability to understand English

Exclusion Criteria:

* A Score of less than 25 on Mini-mental state examination
* Heel bone density with T-score less than <-2.0
* Self-reported metal implants due to any orthopedic conditions
* Presence of any other neurological impairments such as Parkinsons disease, Alzheimers disease, vestibular dysfunction, peripheral neuropathy or unstable epilepsy

Inclusion/Exclusion criteria for Older adults

Inclusion Criteria:

* Participants should be 50 to 90 years of age.
* Able to follow instructions provided in English.
* No history of neurological impairment (Stroke, Parkinson's disease and Multiple Sclerosis).
* Able to stand and walk with or without assistive device or braces as part of their activities of daily living (self-report).
* Cognitive skills to actively participate (score of < 26 on Montreal cognitive assessment indicates cognitive impairment).

Exclusion Criteria:

* Significant cognitive or communicative impairment indicated by a score of > 26 on Montreal cognitive assessment indicates cognitive impairment.
* In neurologically impaired individuals, for cognitive impairment a score of <25 on Mini Mental State Exam Score; for aphasia <71% on Mississippi Aphasia Screening Test and >15 on Geriatric Depression Scale.
* Heel bone density with T-score less than <-2.0
* Participants unavailable for 6 weeks of participation.
* Uncontrolled pain >3/10 on VAS. Complains of shortness of breath.
* Uncontrolled hypertension (systolic blood pressure (SBP) > 165 mmHg and/or diastolic blood pressure (DBP) > 110 mmHg during resting).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2014-12-04 (Actual); Primary Completion 2016-10-25 (Actual); Study Completion 2016-10-25 (Actual)

PRIMARY OUTCOMES:
Change in Movement Velocity (during dual-tasking) | Baseline (Week 0) and Immediate Post-training (Week 7)
  Degrees of movement per second of a self-initiated movement. Higher values indicate better performance.
Change in Postural Stability (during single and dual-tasking) | Baseline (Week 0) and Immediate Post-training (Week 7)
  Postural Stability (Laboratory Slip test) can be defined by simultaneous control of center of mass (COM) position and velocity during slip-like perturbation relative to the rear edge of base of support (rear heel). The position normalized with the individual's foot length, and velocity by square root of gravitational acceleration and individual's body height. Greater values indicate greater stability.
Change Cognitive Accuracy (during dual-tasking) | Baseline (Week 0) and Immediate Post-training (Week 7)
  Accuracy (number of correct responses out of the total responses) during the letter number sequencing task. Higher accuracy indicates better performance.
Compliance to therapy (total time spent over the intervention duration) | Baseline (Week 0) to Post-training (Week 7)
  Compliance will be assessed by logs of participation time (total time summed over the intervention duration). This will assess if participants were able to complete and tolerate the intervention. Higher values indicate more compliance.
Change in reaction time with functional arm reach - Dance therapy for people with stroke and healthy older adults | Baseline (Week 0) and Immediate Post-training (Week 7)
  Reaction time was evaluated with electromyography as the time elapsed between the final cue, "Go" (at 4s), and the onset of EMG signal (calculated as ±1 standard deviation from baseline). Electromyographic will be used to monitor muscle activity in both upper extremities for stand arm reaching. The test will take about 30 minutes.

SECONDARY OUTCOMES:
Change in Berg Balance Scale | Baseline (Week 0) and Immediate Post-training (Week 7)
  Assess static and dynamic balance control. It is a 14 item scale. Score for each item ranges from 0-4. Item score are then summed and maximum score of 54 can be obtained. Less than 45 on this scale indicates a greater risk for falling.
Change in Timed Up and Go test and cognitive Timed up and Go test (seconds) | Baseline (Week 0) and Immediate Post-training (Week 7)
  Assess mobility, balance and walking ability. It is a fall risk predictor. More than 14 seconds taken to complete the test indicates a greater risk for falling.
Change in distance covered in Six minute walk test | Baseline (Week 0) and Immediate Post-training (Week 7)
  Assess endurance and walking ability. Total walking distance covered in 6 minutes was recorded.
Change in performance on Chair Stand Test | Baseline (Week 0) and Immediate Post-training (Week 7)
  Assess balance, functional mobility and strength. It is the number of times the participant completed sit to stand within 30 seconds.
Change in performance on Four Step Square test | Baseline (Week 0) and Immediate Post-training (Week 7)
  Assess balance. The amount of time taken (in seconds) for the participant to complete the sequence of stepping was recorded. More than 15 seconds to complete the test indicates greater risk of falling.
Change in Activity Specific Balance confidence | Baseline (Week 0) and Immediate Post-training (Week 7)
  It is a 16 item self-reported physical activity and community integration questionnaire with each item score ranging from 0-100, where 0 indicates no confidence and 100 indicates complete confidence.
Change in physical activity | Baseline (Week 0) and Immediate Post-training (Week 7)
  For this purpose, the number of steps taken for up to one week will be measured using a wearable sensor by Tractivity (Huston, Texas). During the initial visit, participant will be given the sensor placed in an ankle band. After initial activity monitoring for one week, participants will be scheduled for the training session. After the training participants post-training one-week physical activity will also be monitored. Higher number of steps, indicate more physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Tanvi S Bhatt, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No